CLINICAL TRIAL: NCT06498050
Title: Brolucizumab Efficacy and Safety Single-Arm Descriptive Trial in Patients With Persistent Diabetic Macular Edema
Acronym: BEST
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Beijing Novartis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258BCN03T
Record Dates: First submitted 2024-06-10; First posted 2024-07-12 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; brolucizumab; central subfield thickness; visual acuity; anti-VEGF

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brolucizumab 6mg (Experimental): Brolucizumab 6 mg will be given via intravitreal injections following two treatment patterns: Treatment pattern 1: q6w*5; Treatment pattern 2: q6w*3 +q12w*1
  Interventions: Drug: intravitreal injection of Brolucizumab 6 mg in study eye

INTERVENTIONS:
Drug: intravitreal injection of Brolucizumab 6 mg in study eye — After disinfecting the conjunctival sac and administering a topical anesthetic, an intravitreal injection of Brolucizumab at a dose of 6 mg is given.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of brolucizumab 6 mg in Chinese patients with persistent diabetic macular edema (DME). It will also learn about the safety of brolucizumab 6 mg.

The main questions it aims to answer are:

Does brolucizumab 6 mg reduce central subfield thickness (CST) and improve best-corrected visual acuity (BCVA) of participants? What medical problems do participants have after receiving intravitreal injections of brolucizumab 6 mg? Researchers will compare baseline CST and BCVA to those at each post-baseline visit to see if brolucizumab 6 mg works to treat persistent DME.

Participants will:

Receive brolucizumab 6 mg via intravitreal injections following two treatment patterns:

Treatment Pattern 1: every 6 weeks for 5 injections Treatment Pattern 2: every 6 weeks for 3 injections followed by 1 injection after 12 weeks Visit the clinic 8 times for treatment and assessments over the course of 28 weeks

DETAILED DESCRIPTION:
This study is a single-arm, open-label study designed to evaluate the efficacy and safety of intravitreal injections (IVI) of brolucizumab 6 mg in Chinese subjects with persistent diabetic macular edema (DME). The study consists of a 2-week screening phase, followed by a 28-week period from the point of informed consent.

Intervention, assessments and analyses will be performed in Guangdong Provincial People's Hospital. Data from assessments will be extracted from the patients' medical records at the following time points: baseline, Week 1, Week 6, Week 12, Week 16, Week 18, Week 24, and at Week 28.

Safety data will be collected from any time point thoughout the study. Any adverse events identified will be recorded and treated per recommended standard treatment guideline combined with local clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent had to be obtained prior to participation in the study.
2. Patients ≥18 years of age at screening.
3. Patients with type 1 or type 2 diabetes mellitus and HbA1c of ≤10% at screening.
4. Study Eye: Visual impairment due to DME with: (1) BCVA score between 78 and 23 letters, inclusive, using ETDRS visual acuity testing charts at a starting testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/320) at screening and baseline. (2)DME involving the center of the macula, with central subfield retinal thickness (e.g. measured from retinal pigment epithelium (RPE) to the inner limiting membrane (ILM) inclusively) of ≥320 μm on SD-OCT at screening. (Investigator must verify accuracy of OCT scan by ensuring it is centered and of adequate quality) (3) Media clarity, pupillary dilation, and individual cooperation sufficient for adequate OCTs. (4) Diagnosis of DME less than 6 months prior to enrollment. (5) Have at least 3 intravitreal injections of the same anti-VEGF medication (Ranibizumab, Aflibercept, or Conbercept) within the 20 weeks prior to enrollment.

Exclusion Criteria:

1. Active Proliferative Diabetic Retinopathy in the study eye as per investigator.
2. Concomitant conditions or ocular disorders in the study eye at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention for the duration of the study (e.g. cataract, vitreous hemorrhage, retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause).
3. Any active intraocular or periocular infection or active intraocular inflammation (e.g. infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in study eye at screening or baseline, or any history of intraocular inflammation.
4. Presence of amblyopia, amaurosis or ocular disorders with vision <20/200 (35 letters) in the fellow eye at screening or baseline.
5. History of idiopathic or autoimmune uveitis in the study eye.
6. Any history of intravitreal anti-VEGF treatment in study eye during the 28 days prior to baseline.
7. Use of fluocinolone acetonide intravitreal implant (Iluvien) in study eye at any time. Prior use of other intraocular or periocular corticosteroids in the study eye is not an exclusion provided at least 6-month wash-out prior to baseline.
8. Laser photocoagulation (focal/grid or panretinal) in the study eye during the 3 months prior to baseline.
9. History of vitreoretinal surgery in study eye.
10. Stroke or myocardial infarction during the 6 month period prior to baseline.
11. Any history of renal failure requiring dialysis or kidney transplantation or any history of kidney transplantation.
12. Poor blood pressure control（SBP≥180 mmHg or DBP≥100 mmHg）
13. Any history of systemic anti-VEGF treatment during the 3 months prior to baseline
14. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with central subfield thickness (CST) <300 μm assessed by Spectral Domain Optical Coherence Tomography (SD-OCT) | Baseline, week 28
  Central subfield thickness (CST) will be measured by Spectral Domain Optical Coherence Tomography (SD-OCT). The measurement of CST refers to the mean retinal thickness of the circular area within 1 mm in diameter that centered on the fovea. SD-OCT images will be captured for the study eye using SD-OCT equipment.
The proportion of patients with best-corrected visual acuity (BCVA) improvement of ≥5 letters assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing chartstesting charts | Baseline, week 28
  Best Corrected Visual Acuity (BCVA) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts. Eligible participants will be those with a BCVA ETDRS letter score ranging from 78 to 23 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye. The scoring system for visual function ranges from 0 to 100, with higher score indicating better visual function.

SECONDARY OUTCOMES:
Change in BCVA at each post-baseline visit assessed by ETDRS visual acuity testing charts | Baseline, week 1, week 6, week 12, week 16, week 18, week 24, week 28
  Best Corrected Visual Acuity (BCVA) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts. Eligible participants will be those with a BCVA ETDRS letter score ranging from 78 to 23 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye. The scoring system for visual function ranges from 0 to 100, with higher score indicating better visual function.
The proportion of patients with gain in BCVA of ≥5, ≥10 and ≥15 letters assessed by ETDRS visual acuity testing charts | Baseline, week 28
  Best Corrected Visual Acuity (BCVA) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts. Eligible participants will be those with a BCVA ETDRS letter score ranging from 78 to 23 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye. The scoring system for visual function ranges from 0 to 100, with higher score indicating better visual function.
The proportion of patients with loss in BCVA of ≥5, ≥10 and ≥15 letters assessed by ETDRS visual acuity testing charts | Baseline, week 28
  Best Corrected Visual Acuity (BCVA) was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts. Eligible participants will be those with a BCVA ETDRS letter score ranging from 78 to 23 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye. The scoring system for visual function ranges from 0 to 100, with higher score indicating better visual function.
Change in CST from baseline at each post-baseline visit assessed by SD-OCT | Baseline, week 1, week 6, week 12, week 16, week 18, week 24, week 28
  Central subfield thickness (CST) will be measured by Spectral Domain Optical Coherence Tomography (SD-OCT). The measurement of CST refers to the mean retinal thickness of the circular area within 1 mm in diameter that centered on the fovea. SD-OCT images will be captured for the study eye using SD-OCT equipment.
The proportion of patients with CST <280 μm assessed by SD-OCT at each post-baseline visit | Baseline, week 1, week 6, week 12, week 16, week 18, week 24, week 28
  Central subfield thickness (CST) will be measured by Spectral Domain Optical Coherence Tomography (SD-OCT). The measurement of CST refers to the mean retinal thickness of the circular area within 1 mm in diameter that centered on the fovea. SD-OCT images will be captured for the study eye using SD-OCT equipment.
The proportion of patients with presence of subretinal fluid (SRF), intraretinal fluid (IRF) and simultaneous absence of SRF and IRF at each post-baseline visit assessed by SD-OCT | Baseline, week 1, week 6, week 12, week 16, week 18, week 24, week 28
  Subretinal Fluid (SRF) and Intraretinal Fluid (IRF) will be evaluated in images captured for the study eye using SD-OCT equipment.
Change in SRF and IRF from baseline assessed by quantitative criteria based on SD-OCT | Baseline, week 28
  The volume of SRF and IRF will be calculated in SD-OCT images using artificial intelligence algorithms.
Change in vessel densities of deep capillary plexus (DCP), superficial capillary plexus (SCP) and radial peripapillary capillaries (RPC), and foveal avascular zone (FAZ) area from baseline based on optical coherence tomography angiography (OCTA) | Baseline, week 28
  Optical coherence tomography-angiography (OCT-A) is a dye-less and non-invasive angiographic technique that offers a three-dimension imaging of the retinal circulation. It enables visualizing the movement of particles within blood vessels, predominantly red blood cells, across the entire retinal and choroidal vascular layers.
The proportion of patients with a ≥2- and ≥3-step improvement or worsening from baseline assessed by the ETDRS Diabetic Retinopathy Severity Scale (DRSS) score | Baseline, week 28
  The Early Treatment Diabetic Retinopathy Study Diabetic Retinopathy Severity Scale (DRSS) is a standard approach to measure diabetic retinopathy (DR) severity. Wide-field fundus color photography images were obtained and assessed in the study eye by fundus color photography machines.
The proportion of patients with presence of leakage assessed by qualitative and quantitative criteria based on ultrawide-field fluorescein angiography (UWFFA) | Baseline, week 28
  Fluorescein Angiography (FA) is an invasive eye examination that uses an injected dye to illuminate the retinal and choroidal blood vessels, offering a dynamic, real-time assessment of blood flow and leakage
The proportions of patients treated with 4 and 5 injections | Baseline, week 28
  There are 2 treatment patterns depending on the disease activity assessment at week 18. Treatment Pattern 1: every 6 weeks for 5 injections; Treatment Pattern 2: every 6 weeks for 3 injections followed by 1 injection after 12 weeks.
Incidence and characteristics of ocular and non-ocular adverse events | Baseline, week 28
  An adverse event is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings, symptom or disease) in a clinical investigation The ocular adverse events will be assessed by slip-lamp examination, intraocular pressure from non-contact tonometry, and retinal circulation from optical coherence tomography angiography. The non-ocular adverse events will be assessed by vital signs, complete blood count, biochemical profile, glycosylated hemoglobin A1c, urinary albumin to creatinine ratio, serum pregnancy test, and urine pregnancy test.

OTHER OUTCOMES:
Change in aqueous cytokine levels assessed by immunological methods from baseline | immediately before the first injection at week 1, immediately before the last injection at week 24
  The cytokines detected in aqueous humor will be quantitatively assessed by immunological methods.
Longitudinal changes of leakage in UWFFA | Baseline, week 28
  Fluorescein Angiography (FA) is an invasive eye examination that uses an injected dye to illuminate the retinal and choroidal blood vessels, offering a dynamic, real-time assessment of blood flow and leakage.
Imaging predictors in SD-OCT: disorganization of retinal inner layers (DRIL), hyperreflective foci (HRF), integrity of the ellipsoid zone (EZ), IRF volume, SRF volume | Baseline, week 28
  Disorganization of retinal inner layers (DRIL), hyperreflective foci (HRF), integrity of the ellipsoid zone (EZ), IRF volume, SRF volume will be evaluated in images captured for the study eye using SD-OCT equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Honghua Yu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Hu Y, Shen C, Li J, Liang A, Fang Y, Zeng J, Liao H, Zheng C, Ouyang S, Hu Y, Cao D, Yu H. Brolucizumab efficacy and safety single-arm descriptive trial in patients with persistent diabetic macular edema (BEST study): protocol for a single-centre, open-label, single-arm clinical trial in China. BMJ Open. 2025 Jul 28;15(7):e099551. doi: 10.1136/bmjopen-2025-099551. PMID 40721260